CLINICAL TRIAL: NCT00593697
Title: A Randomized Phase III Study Comparing Trastuzumab Plus Docetaxel (HT) Followed by 5-FU, Epirubicin, and Cyclophosphamide (FEC) to the Same Regimen Followed by Single-agent Trastuzumab as Adjuvant Treatments for Early Breast Cancer
Brief Title: The Synergism Or Long Duration (SOLD) Study
Acronym: SOLD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Finnish Breast Cancer Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Protocol number FBCSG-01-2007; EudraCT number 2007-002016-26
Record Dates: First submitted 2008-01-03; First posted 2008-01-15 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Breast Neoplasms
Keywords: breast cancer; adjuvant therapy; trastuzumab; chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Docetaxel; CEF regimen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Weekly or 3-weekly trastuzumab plus 3-weekly docetaxel (3 cycles) (HT) -> 3-weekly FE75C (3 cycles) (HT x3 -> FE75C x3)
  Interventions: Drug: trastuzumab (9 weeks) + docetaxel
- B (Active Comparator): Weekly or 3-weekly trastuzumab plus 3-weekly docetaxel (3 cycles) (HT) -> 3-weekly FE75C (3 cycles) -> trastuzumab to complete 1 year (14 3-weekly infusions) (HT x3 ->FE75C x3 -> H3wkly x14)
  Interventions: Drug: trastuzumab (9 weeks) + docetaxel + CEF + trastuzumab (up to 51 weeks)

INTERVENTIONS:
Drug: trastuzumab (9 weeks) + docetaxel — Patients diagnosed with early breast cancer with a high risk of disease recurrence will be randomly allocated to one of the following 2 arms in a 1:1 ratio:
  A. Weekly or 3-weekly trastuzumab plus 3-weekly docetaxel (3 cycles) (HT) -> 3-weekly FE75C (3 cycles) (HT x3 ->FE75C x3) B. Weekly or 3-weekly trastuzumab plus 3-weekly docetaxel (3 cycles) (HT) -> 3-weekly FE75C (3 cycles) -> trastuzumab to complete 1 year (14 3-weekly infusions) (HT x3 ->FE75C x3 -> H3wkly x14)
  Arms: A
Drug: trastuzumab (9 weeks) + docetaxel + CEF + trastuzumab (up to 51 weeks) — Weekly or 3-weekly trastuzumab plus 3-weekly docetaxel (3 cycles) (HT) -> 3-weekly FE75C (3 cycles) -> trastuzumab to complete 1 year (14 3-weekly infusions) (HT x3 ->FE75C x3 -> H3wkly x14)
  Arms: B

SUMMARY:
The purpose of the study is to compare disease-free survival (DFS) of women treated with concomitant trastuzumab plus docetaxel followed by FEC to that of the women treated with the same regimen followed by single-agent trastuzumab to complete one year of trastuzumab administration as adjuvant treatments of early HER2-positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has provided a written informed consent prior to study-specific screening procedures, with the understanding that she has the right to withdraw from the study at any time, without prejudice.
2. Woman > 18 years of age.
3. Histologically confirmed invasive breast cancer.
4. HER2-positive breast cancer (preferably assessed with CISH or FISH; if not available with immunohistochemistry 3+)
5. A high risk of breast cancer recurrence with one of the following:

   * Pathological N0 with the longest invasive tumor diameter >5 mm
   * Histologically confirmed regional node positive disease (pN+; nodal isolated tumor cells/cell clusters < 0.2 mm in diameter (ITP) are not counted as a metastasis)

Exclusion Criteria:

1. Presence of distant metastases.
2. Inflammatory breast cancer.
3. pT1bN0M0 (i.e. the longest tumor diameter 6 to 10 mm, node-negative) and histological grade 1.
4. Clinically significant (i.e. active) cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmia not well controlled with medication) or myocardial infarction within the last 12 months.
5. Left ventricular ejection fraction less than 50% (or under the institutional normal reference range) assessed by echocardiography or isotope cardiography.
6. ER, PgR and HER-2 status (via in situ hybridization or immunohistochemistry) not determined.
7. Primary systemic cancer therapy (neoadjuvant chemotherapy or endocrine therapy) has been administered prior to breast surgery.
8. The WHO performance status > 1.
9. Pregnant or lactating women.
10. Women of childbearing potential unless using a reliable and appropriate contraceptive method. Women must have been amenorrheic for at least 12 months prior to study entry to be considered postmenopausal and to have no childbearing potential. Women of childbearing potential (menstruating within 12 months of study entry), or with no hysterectomy and age < 55, must have a negative pregnancy test at baseline.
11. More than 12 weeks between breast surgery and date of randomization.
12. Organ allografts with immunosuppressive therapy required.
13. Major surgery (except breast surgery) within 4 weeks prior to study treatment start, or lack of complete recovery from the effects of major surgery.
14. Participation in any investigational drug study within 4 weeks preceding treatment start.
15. Patients with a history of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant precluding study participation.
16. History of another malignancy within the last five years except cured basal cell carcinoma of skin or carcinoma in situ of the uterine cervix.
17. One or more of the following:

    * Blood hemoglobin < 10.0 g/dL, neutrophils < 1.5 x 109/L, platelet count < 120 x 109/L
    * Serum/plasma creatinine > 1.5 x Upper Limit of Normal (ULN)
    * Serum/plasma bilirubin > ULN
    * Serum/plasma ALT and/or AST > 1.5 x ULN
    * Serum/plasma alkaline phosphatase > 2.5 x ULN
18. Serious uncontrolled infection or other serious uncontrolled concomitant disease.
19. Unwilling or unable to comply with the protocol for the duration of the study.
20. History of hypersensitivity to the investigational products or to drugs with similar chemical structures.
21. Pre-existing motor or sensory neurotoxicity of a severity ≥ grade 2 by CTCAE version 3, unless related to mechanical etiology.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2168 (Actual)
Dates: Start 2008-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | 3-10years

SECONDARY OUTCOMES:
Overall survival, distant disease-free survival, cardiac event-free disease-free survival, left ventricle ejection fractions, adverse events, quality of life | 3-10years

CONTACTS AND LOCATIONS:
Locations (1):
- Helsinki University Central Hospital, Department of Oncology, Helsinki, Finland

REFERENCES:
- [Derived] Joensuu H, Fraser J, Wildiers H, Huovinen R, Auvinen P, Utriainen M, Villman KK, Halonen P, Granstam-Bjorneklett H, Tanner M, Sailas L, Turpeenniemi-Hujanen T, Yachnin J, Huttunen T, Neven P, Canney P, Harvey VJ, Kellokumpu-Lehtinen PL, Lindman H. Long-Term Outcomes of Adjuvant Trastuzumab for 9 Weeks or 1 Year for ERBB2-Positive Breast Cancer: A Secondary Analysis of the SOLD Randomized Clinical Trial. JAMA Netw Open. 2024 Aug 1;7(8):e2429772. doi: 10.1001/jamanetworkopen.2024.29772. PMID 39186271
- [Derived] Joensuu H, Fraser J, Wildiers H, Huovinen R, Auvinen P, Utriainen M, Nyandoto P, Villman KK, Halonen P, Granstam-Bjorneklett H, Lundgren L, Sailas L, Turpeenniemi-Hujanen T, Tanner M, Yachnin J, Ritchie D, Johansson O, Huttunen T, Neven P, Canney P, Harvey VJ, Kellokumpu-Lehtinen PL, Lindman H. Effect of Adjuvant Trastuzumab for a Duration of 9 Weeks vs 1 Year With Concomitant Chemotherapy for Early Human Epidermal Growth Factor Receptor 2-Positive Breast Cancer: The SOLD Randomized Clinical Trial. JAMA Oncol. 2018 Sep 1;4(9):1199-1206. doi: 10.1001/jamaoncol.2018.1380. PMID 29852043